CLINICAL TRIAL: NCT00064714
Title: Effect of AC 2993 (Synthetic Exendin-4) - Administered Alone or in Combination With Daclizumab - on Islet Function in Patients With Type I Diabetes
Brief Title: Effect of AC2993 With or Without Immunosuppression on Beta Cell Function in Patients With Type I Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 030245 (2993T1-101); 03-DK-0245
Record Dates: First submitted 2003-07-10; First posted 2003-07-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus (T1DM); Beta-Cell; C-Peptide; Immunosuppression; Insulin; Islet; Function; AC2993 (Synthetic Exendin-4); Diabetes Mellitus; Type I Diabetes Mellitus; T1DM
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Exenatide; Daclizumab; Immunosuppressive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): Group 1 will receive immunosuppression and AC2993; then immunosuppression only
  Interventions: Drug: AC2993 (exenatide); Drug: daclizumab (immunosuppressive)
- Group 2 (Experimental): Group 2 will receive AC2993 only; then neither immunosuppression nor AC2993
  Interventions: Drug: AC2993 (exenatide); Drug: daclizumab (immunosuppressive)
- Group 3 (Experimental): Group 3 will receive immunosuppression and AC2993; then immunosuppression and AC2993
  Interventions: Drug: AC2993 (exenatide); Drug: daclizumab (immunosuppressive)
- Group 4 (Experimental): Group 4 will receive AC2993 only; then AC2993 only
  Interventions: Drug: AC2993 (exenatide); Drug: daclizumab (immunosuppressive)

INTERVENTIONS:
Drug: AC2993 (exenatide) — Dose-escalation beginning with 2.5 μg administered subcutaneously twice per day (BID); then to 2.5 μg four times a day (QID); then to 5 μg four times a day; then to 10 μg four times a day.
Drug: daclizumab (immunosuppressive) — 2 mg/kg intravenously infused over 30 minutes every month for 12 months

SUMMARY:
This study will determine 1) the safety of AC2993 in patients with type I diabetes; 2) the ability of AC2993 to improve beta cell function; and 3) the effects of immunosuppression on beta cell function.

Type I diabetes is an autoimmune disease, in which the immune system attacks the beta cells of the pancreas. These cells produce insulin, which regulates blood sugar. AC2993 may improve the pancreas's ability to produce insulin and help control blood sugar, but it may also activate the original immune response that caused the diabetes. Thus, this study will examine the effects of AC2993 alone as well as in combination with immunosuppressive drugs.

Patients between 18 and 60 years of age who have type I diabetes mellitus may be eligible for this 20-month study. They must have had diabetes for at least 5 years and require insulin treatment. Candidates will be screened with a questionnaire, followed by medical history and physical examination, blood and urine tests, a chest x-ray and skin test for tuberculosis, electrocardiogram (EKG), and arginine stimulated C-peptide test (see description below). Participants will undergo the following tests and procedures:

Advanced screening phase: Participants undergo a diabetes education program, including instruction on frequent blood glucose monitoring, dietary education on counting carbohydrates, intensive insulin therapy, review of signs and symptoms of low blood sugar (hypoglycemia), and potential treatment with glucagon shots.

Patients must administer insulin via an insulin pump or take at least four injections per day including glargine (Lantus) insulin.

4-month run-in phase

* Arginine-stimulated C-peptide test: This test measures the body's insulin production. The patient is injected with a liquid containing arginine, a normal constituent of food that increases insulin release from beta cells into the blood stream. After the injection, seven blood samples are collected over 10 minutes.
* Mixed meal stimulated C-peptide test with acetaminophen: This test assesses the response of the beta cells to an ordinary meal and the time it takes for food to pass through the stomach. The patient drinks a food supplement and takes acetaminophen (Tylenol). Blood samples are then drawn through a catheter (plastic tube placed in a vein) every 30 minutes for 4 hours to measure levels of various hormones and the concentration of acetaminophen.
* Euglycemic clamp: This test measures the body's level of insulin resistance by measuring the amount of glucose necessary to compensate for an increased insulin level while maintaining a prespecified blood glucose level.

DETAILED DESCRIPTION:
Type I diabetes mellitus (T1DM) typically results from immune mediated destruction of pancreatic beta cells. Previous studies indicate that some patients retain the capacity for limited endogenous insulin production. AC2993 (synthetic exendin-4) has been shown in preclinical and in human studies to have several potentially beneficial antidiabetic actions, including recovery and neogenesis of pancreatic islets. Thus, we plan to enroll adults with long-standing T1DM who have some C-peptide secretion indicating residual beta cell mass. The latter will be targeted by AC2993. Due to the possibility of stimulating the underlying autoimmune process of T1DM, especially if islet regeneration occurs, we will subject half of the enrollees to immunosuppression. We plan to study the effects of AC2993 alone, immunosuppression (daclizumab) alone, as well as the combination of AC2993 and immunosuppression on insulin secretion and glycemia control.

ELIGIBILITY:
* INCLUSION CRITERIA:

T1DM for at least 5 years as defined by the following:

1. Insulin dependence (with an insulin requirement less than 0.8 units/kg/day).
2. Current or past anti-islet antibodies (anti-insulin before initiation of insulin therapy, anti-islet cell (ICA), anti-tyrosine phosphatase IA-2, and/or anti-glutamic acid decarboxylase (GAD65) antibodies).
3. BMI greater than or equal to 20 kg/m(2) and less than or equal to 30 kg/m(2).

C-peptide greater than or equal to 0.3 and less than or equal to 1.2 ng/mL at baseline or during an arginine-stimulated C-peptide test.

Age 18 to 60 years, inclusive.

EXCLUSION CRITERIA:

Symptomatic gastroparesis.

Diabetic nephropathy with a creatinine clearance less than 60 cc/min or 24-hour urine albumin greater than 300 mg.

Insulin requirements greater than 0.8 units/kg/day.

Hypoglycemia unawareness: Unless easily corrected via simple modifications in the patient's diabetes regimen, the potential enrollee will be excluded if he/she has suffered greater than or equal to 2 episodes of severe hypoglycemia during the most recent 12 months, defined as requiring assistance from a third party, receiving assistance from medics, visiting an ER or being hospitalized due to the hypoglycemia.

Evidence of chronic infection.

History of any malignancy.

Any chronic medical condition that unduly increase risk for the potential enrollee as judged by study investigators.

Hematologic abnormalities:

1. Anemia (hematocrit less than 31.8% in women and less than 36.7% in men).
2. Leukopenia (WBC count less than 3.4 K/mm(3)).
3. Thrombocytopenia (platelet count less than 162 K/mm(3)).

Hypertension, whether untreated or resistant to medical treatment, with blood pressure greater than 140/85 mm Hg.

Pregnancy, breastfeeding or planned pregnancy within two years.

Unable to identify primary care provider willing to partner with study investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2003-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change in basal C-peptide level | baseline and 6 months
  Assess whether patients treated with AC2993 (with or without concomitant immunosuppression) will display at least a 50% improvement in their basal C-peptide level. C-peptide level is a surrogate measure for insulin production.

CONTACTS AND LOCATIONS:
Overall Officials: Vice President, Research and Development, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bach JF, Chatenoud L. Tolerance to islet autoantigens in type 1 diabetes. Annu Rev Immunol. 2001;19:131-61. doi: 10.1146/annurev.immunol.19.1.131. PMID 11244033
- [Background] Lernmark A, Barmeier H, Dube S, Hagopian W, Karlsen A, Wassmuth R. Autoimmunity of diabetes. Endocrinol Metab Clin North Am. 1991 Sep;20(3):589-617. PMID 1935920
- [Background] Mathis D, Vence L, Benoist C. beta-Cell death during progression to diabetes. Nature. 2001 Dec 13;414(6865):792-8. doi: 10.1038/414792a. PMID 11742411
- [Derived] Rother KI, Spain LM, Wesley RA, Digon BJ 3rd, Baron A, Chen K, Nelson P, Dosch HM, Palmer JP, Brooks-Worrell B, Ring M, Harlan DM. Effects of exenatide alone and in combination with daclizumab on beta-cell function in long-standing type 1 diabetes. Diabetes Care. 2009 Dec;32(12):2251-7. doi: 10.2337/dc09-0773. Epub 2009 Oct 6. PMID 19808924
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2003-DK-0245.html